CLINICAL TRIAL: NCT06715098
Title: Comparison of Robot Assisted Gait Training and Body Weight Supported Treadmill Training in Chronic Stroke Patients Using Gait Analysis and SEMG Measurements
Brief Title: Comparison of Robot Assisted Gait Training and Body Weight Supported Treadmill Training Using Gait Analysis and SEMG Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Füsun Ardıç, Professor Doctor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PamukkaleU.ftr-FArdıç-001
Record Dates: First submitted 2024-07-12; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Stroke, Ischemic
Keywords: Stroke; RehaWalk; RoboGait
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RoboGait group (Experimental): Robotic walking training 3 days a week, 30 minutes a day for 4 weeks
  Interventions: Device: RoboGait
- RehaWalk group (Experimental): Walking training on treadmill with body weight support for 30 minutes a day, 3 days a week for 4 weeks
  Interventions: Device: RehaWalk
- Conventional Group (Active Comparator): Conventional walking training for 30 minutes a day, 3 days a week for 4 weeks
  Interventions: Other: Conventional

INTERVENTIONS:
Device: RoboGait — RoboGait: robotic-assisted gait training
  Arms: RoboGait group
Device: RehaWalk — RehaWalk: body weight-supported treadmill training
  Arms: RehaWalk group
Other: Conventional — Conventional: conventional walking training
  Arms: Conventional Group

SUMMARY:
The aim of our randomized controlled clinical trial was to analyze the effects of robotic-assisted gait training and body-weight-supported treadmill training on gait analysis parameters and lower extremity agonist and antagonist muscle activities in stroke patients and to compare their effectiveness in improving locomotor function. The main questions that the researchers aimed to answer are: What are the effects of robotic-assisted gait training and body-weight-supported treadmill training on gait analysis parameters in stroke patients? What are the effects of robotic-assisted gait training and body-weight-supported treadmill training on lower extremity agonist and antagonist muscle activities in stroke patients? What is the effectiveness of robotic-assisted gait training and body-weight-supported treadmill training in improving locomotor function in stroke patients? The patients included in the study were randomly divided into three groups: The first group received robotic-assisted gait training with RoboGait, the second group received body-weight-supported gait training on a treadmill with RehaWalk, and the third group received conventional walking training.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Chronic stage stroke (6 months - 2 years)
* First stroke
* Spasticity of Ashworth stage 2 or lower
* Ability to follow commands
* Ability to walk unsupported for more than 10 meters
* No treatment received in the last month

Exclusion Criteria:

* Severe osteoporosis
* Unstable fracture
* Excessive spasticity (Ashworth stage 3 and above)
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Gait analysis with 2D camera | Change from baseline kinematic parameters at the 4th week after the treatment
  Kinematic parameters: Hip joint flexion range of motion degree in the swing phase in the sagittal plane, knee joint maximum flexion angle degree, ankle joint dorsiflexion range of motion degree
Surface Electromyography (sEMG) | Change from baseline surface electromyography (sEMG) at the 4th week after the treatment
  The average EMG (AEMG) amplitude and co-contraction indices (CCI) are calculated for the affected lower extremity's knee flexion and ankle dorsiflexion during the swing phase. CCI is calculated using the formula antagonistic muscle AEMG / (antagonistic muscle AEMG + agonistic muscle AEMG)
Pressure and Walking Analysis | Change from baseline pressure and walking analysis at the 4th week after the treatment
  The researchers examined the effects such as walking line length, single support line, forward and backward rollers and lateral symmetry indexes in the pressure analyses. In the gait analysis, walking speed, cadence, step length, step width, foot rotation angle, step duration, double support duration, stance phase, swing phase, single support phase, pre-swing phase, mid-swing phase, terminal swing phase, stance duration, swing duration, double phase, double step length and temporal symmetry index were evaluated. The temporal symmetry index was calculated using the following formula: Swing duration of the affected side of the patient / Swing duration of the unaffected side of the patient

SECONDARY OUTCOMES:
The Functional Ambulation Scale (FAS) | Change from baseline FAS at the 4th week after the treatment
  The Functional Ambulation Scale (FAS) is a scale used to assess the level of ambulation in patients. It is divided into six categories graded from 0 to 5: FAS 0: no ambulation, FAS 1-2: unable to walk without assistance, FAS 3-5: able to walk 6 meters independently.
For lower extremity, the Fugl-Meyer Assessment (FMA-LE) | Change from baseline FMA-LE at the 4th week after the treatment
  For lower extremity, the Fugl-Meyer Assessment (FMA-LE) was used in our study, consisting of a total of 17 items with a maximum score of 34 points. The scale assesses reflexes, synergy-dependent or synergy-independent voluntary movements, coordination, and speed. Each item is scored between 0 and 2 points, with a higher score indicating better outcomes.
The 6-minute walk test (6MWT) | Change from baseline 6MWT at the 4th week after the treatment
  In the 6-minute walk test (6MWT), researchers asked participants to walk down a 30-meter hospital hallway at their own pace for 6 minutes, following standard instructions to cover as much distance as possible. The distance walked was recorded in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Füsun Ardıç, Professor, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuriakose D, Xiao Z. Pathophysiology and Treatment of Stroke: Present Status and Future Perspectives. Int J Mol Sci. 2020 Oct 15;21(20):7609. doi: 10.3390/ijms21207609. PMID 33076218
- [Background] GBD 2016 Stroke Collaborators. Global, regional, and national burden of stroke, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):439-458. doi: 10.1016/S1474-4422(19)30034-1. Epub 2019 Mar 11. PMID 30871944
- [Background] Stroke, Cerebrovascular accident, WHO. Accessed: 08.10.2023 https://www.emro.who.int/health-topics/stroke-cerebrovascular-accident/index.html
- [Background] Furie K. Epidemiology and Primary Prevention of Stroke. Continuum (Minneap Minn). 2020 Apr;26(2):260-267. doi: 10.1212/CON.0000000000000831. PMID 32224751
- [Background] Buntin MB, Colla CH, Deb P, Sood N, Escarce JJ. Medicare spending and outcomes after postacute care for stroke and hip fracture. Med Care. 2010 Sep;48(9):776-84. doi: 10.1097/MLR.0b013e3181e359df. PMID 20706167
- [Background] Selves C, Stoquart G, Lejeune T. Gait rehabilitation after stroke: review of the evidence of predictors, clinical outcomes and timing for interventions. Acta Neurol Belg. 2020 Aug;120(4):783-790. doi: 10.1007/s13760-020-01320-7. Epub 2020 Mar 12. PMID 32166723
- [Background] Druzbicki M, Przysada G, Guzik A, Brzozowska-Magon A, Kolodziej K, Wolan-Nieroda A, Majewska J, Kwolek A. The Efficacy of Gait Training Using a Body Weight Support Treadmill and Visual Biofeedback in Patients with Subacute Stroke: A Randomized Controlled Trial. Biomed Res Int. 2018 Apr 5;2018:3812602. doi: 10.1155/2018/3812602. eCollection 2018. PMID 29850509
- [Background] Malik AN, Tariq H, Afridi A, Rathore FA. Technological advancements in stroke rehabilitation. J Pak Med Assoc. 2022 Aug;72(8):1672-1674. doi: 10.47391/JPMA.22-90. PMID 36280946
- [Background] Norouzi-Gheidari N, Archambault PS, Fung J. Effects of robot-assisted therapy on stroke rehabilitation in upper limbs: systematic review and meta-analysis of the literature. J Rehabil Res Dev. 2012;49(4):479-96. doi: 10.1682/jrrd.2010.10.0210. PMID 22773253
- [Background] Schwartz I, Meiner Z. Robotic-assisted gait training in neurological patients: who may benefit? Ann Biomed Eng. 2015 May;43(5):1260-9. doi: 10.1007/s10439-015-1283-x. Epub 2015 Feb 28. PMID 25724733
- [Background] Yoo HJ, Bae CR, Jeong H, Ko MH, Kang YK, Pyun SB. Clinical efficacy of overground powered exoskeleton for gait training in patients with subacute stroke: A randomized controlled pilot trial. Medicine (Baltimore). 2023 Jan 27;102(4):e32761. doi: 10.1097/MD.0000000000032761. PMID 36705351
- [Background] Özbudak Demir S. Robot-Assisted Gait Training for Patients with Spinal Cord Injury. Turk J Phys Med Rehab 2015;61 (Supp. 1):S37-S44.
- [Background] Visintin M, Barbeau H, Korner-Bitensky N, Mayo NE. A new approach to retrain gait in stroke patients through body weight support and treadmill stimulation. Stroke. 1998 Jun;29(6):1122-8. doi: 10.1161/01.str.29.6.1122. PMID 9626282
- [Background] Zhang H, Li X, Gong Y, Wu J, Chen J, Chen W, Pei Z, Zhang W, Dai L, Shu X, Shen C. Three-Dimensional Gait Analysis and sEMG Measures for Robotic-Assisted Gait Training in Subacute Stroke: A Randomized Controlled Trial. Biomed Res Int. 2023 Apr 11;2023:7563802. doi: 10.1155/2023/7563802. eCollection 2023. PMID 37082189
- [Background] Lura DJ, Venglar MC, van Duijn AJ, Csavina KR. Body weight supported treadmill vs. overground gait training for acute stroke gait rehabilitation. Int J Rehabil Res. 2019 Sep;42(3):270-274. doi: 10.1097/MRR.0000000000000357. PMID 31094879
- [Background] Middleton A, Merlo-Rains A, Peters DM, Greene JV, Blanck EL, Moran R, Fritz SL. Body weight-supported treadmill training is no better than overground training for individuals with chronic stroke: a randomized controlled trial. Top Stroke Rehabil. 2014 Nov-Dec;21(6):462-76. doi: 10.1310/tsr2106-462. PMID 25467394
- [Background] Mao YR, Lo WL, Lin Q, Li L, Xiao X, Raghavan P, Huang DF. The Effect of Body Weight Support Treadmill Training on Gait Recovery, Proximal Lower Limb Motor Pattern, and Balance in Patients with Subacute Stroke. Biomed Res Int. 2015;2015:175719. doi: 10.1155/2015/175719. Epub 2015 Nov 16. PMID 26649295
- [Background] Choi W. Effects of Robot-Assisted Gait Training with Body Weight Support on Gait and Balance in Stroke Patients. Int J Environ Res Public Health. 2022 May 10;19(10):5814. doi: 10.3390/ijerph19105814. PMID 35627346
- [Background] Tanaka N, Yano H, Ebata Y, Ebihara K. Influence of Robot-Assisted Gait Training on Lower-Limb Muscle Activity in Patients With Stroke: Comparison With Conventional Gait Training. Ann Rehabil Med. 2023 Jun;47(3):205-213. doi: 10.5535/arm.22147. Epub 2023 Jun 8. PMID 37317795
- [Background] Brunelli S, Iosa M, Fusco FR, Pirri C, Di Giunta C, Foti C, Traballesi M. Early body weight-supported overground walking training in patients with stroke in subacute phase compared to conventional physiotherapy: a randomized controlled pilot study. Int J Rehabil Res. 2019 Dec;42(4):309-315. doi: 10.1097/MRR.0000000000000363. PMID 31425349
- [Background] Esquenazi A, Lee S, Wikoff A, Packel A, Toczylowski T, Feeley J. A Comparison of Locomotor Therapy Interventions: Partial-Body Weight-Supported Treadmill, Lokomat, and G-EO Training in People With Traumatic Brain Injury. PM R. 2017 Sep;9(9):839-846. doi: 10.1016/j.pmrj.2016.12.010. Epub 2017 Jan 16. PMID 28093370
- [Background] Lee JH, Lee MH. The effects of smartphone multitasking on gait and dynamic balance. J Phys Ther Sci. 2018 Feb;30(2):293-296. doi: 10.1589/jpts.30.293. Epub 2018 Feb 28. PMID 29545698
- [Background] Holden MK, Gill KM, Magliozzi MR, Nathan J, Piehl-Baker L. Clinical gait assessment in the neurologically impaired. Reliability and meaningfulness. Phys Ther. 1984 Jan;64(1):35-40. doi: 10.1093/ptj/64.1.35. PMID 6691052
- [Background] Sullivan KJ, Tilson JK, Cen SY, Rose DK, Hershberg J, Correa A, Gallichio J, McLeod M, Moore C, Wu SS, Duncan PW. Fugl-Meyer assessment of sensorimotor function after stroke: standardized training procedure for clinical practice and clinical trials. Stroke. 2011 Feb;42(2):427-32. doi: 10.1161/STROKEAHA.110.592766. Epub 2010 Dec 16. PMID 21164120
- [Background] Warutkar V, Dadgal R, Mangulkar UR. Use of Robotics in Gait Rehabilitation Following Stroke: A Review. Cureus. 2022 Nov 4;14(11):e31075. doi: 10.7759/cureus.31075. eCollection 2022 Nov. PMID 36475123
- [Background] Lefeber N, De Keersmaecker E, Henderix S, Michielsen M, Kerckhofs E, Swinnen E. Physiological Responses and Perceived Exertion During Robot-Assisted and Body Weight-Supported Gait After Stroke. Neurorehabil Neural Repair. 2018 Dec;32(12):1043-1054. doi: 10.1177/1545968318810810. Epub 2018 Nov 12. PMID 30417724
- [Background] RehaWalk - Ganganalyse und Training. Erişim: 08.10.2023 https://www.zebris.de/medizin/rehawalkr-ganganalyse-und-gangtraining-in-der-rehabilitation.
- [Background] Bedla M, Pieta P, Kaczmarski D, Deniziak S. Estimation of Gross Motor Functions in Children with Cerebral Palsy Using Zebris FDM-T Treadmill. J Clin Med. 2022 Feb 12;11(4):954. doi: 10.3390/jcm11040954. PMID 35207227
- [Background] Yang YR, Chen IH, Liao KK, Huang CC, Wang RY. Cortical reorganization induced by body weight-supported treadmill training in patients with hemiparesis of different stroke durations. Arch Phys Med Rehabil. 2010 Apr;91(4):513-8. doi: 10.1016/j.apmr.2009.11.021. PMID 20382280